CLINICAL TRIAL: NCT01762397
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Dose-escalation Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetics, and Food Effect of PMK-S005 After Oral Administration in Healthy Male Volunteers
Brief Title: A Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetics, and Food Effect of PMK-S005 After Oral Administration in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMK-S005
Record Dates: First submitted 2012-12-20; First posted 2013-01-07 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Gastritis; Gastric Ulcer
MeSH Terms: conditions — Gastritis; Stomach Ulcer | interventions — PMK-S005

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- PMK-S005 (Experimental)
  Interventions: Drug: PMK-S005

INTERVENTIONS:
Drug: PMK-S005

SUMMARY:
The Purpose of a randomized, double-blind, placebo-controlled, single-dose, dose-escalation clinical trial is to explore investigate the safety, tolerability, pharmacokinetics, and food effect of PMK-S005 after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male 20 year ≤ age ≤ 40 year.
* Weight ≥ 55kg, IBW ±20%.
* Patients with normal hematology, biochemistry, urinary result.
* Patients who have not congenital or chronic disease.
* Provision of written informed consent voluntarily.

Exclusion Criteria:

* Patients having known hypersensitivity to any component of the study drug.
* Patients with a history of abnormal digestive organ, kidney, respiratory, neuroendocrine, cardiovascular, hemato-oncology, urinary, muscloskeletal, immune, the nose and ears, psychiatry, stomach system.
* Patients with any gastrointestinal disorders.
* Systolic blood pressure ≥ 150 or ≤ 90 mmHg, Diasolic blood pressure ≥ 95 or ≤ 50 mmHg.
* Drug abuser, alcoholic.
* Patients taking ETC medication within 14 days, OTC within 7 days.
* Patients taking other investigational product within 60 days prior to the participation in the study.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety | 8day
  1. Adverse Event: symptom, start day and time, end day and time, injection time, severity, progress, outcome, relation with investigational product.
  2. Before and after physical examination
  3. Before and after bital Sign: blood pressure, pulse rate, temperature.
  4. Before and after 12-ECG: ventricular rate (/min), PR interval (msec), QRS duration (msec), QT/QTc interval (msec.
  5. Lab: hematologic examination, blood coagulation examination,urine examination
Pharmacokinetics | 8day
  1. Blood evaluation variables: Cmax, AUCt (t=48 h), AUC∞, tmax, CL/F, t1/2.
  2. Urine evaluation variables: Aet (t=48 h), Ae∞, urine recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam national university hospital, Daejeon, Chungcheongnam-do, South Korea